CLINICAL TRIAL: NCT04101032
Title: eBEfree - an ICT Adaptation of BEfree: an APP Delivered Programme Based on Mindfulness, Values, and Compassion for Binge Eating
Brief Title: eBEfree - an ICT Adaptation of BEfree
Acronym: eBEfree
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, José Augusto Pinto Gouveia, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eBEfree; POCI-01-0145-FEDER-029081 (Other Grant/Funding Number: FCT)
Record Dates: First submitted 2019-07-26; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Binge-Eating Disorder
Keywords: Mindfulness; Self-compassion; Values; Binge Eating
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eBEfree (Experimental): eBEfree is a ICT-delivery version of BEfree - eBEfree that comprises 12 online sessions, based on mindfulness,values and compassion components for women with Binge Eating.
  Interventions: Behavioral: eBEfree
- Waiting List (No Intervention): Participants will remain in a waiting list. After 12 weeks, they will be offered the same intervention.

INTERVENTIONS:
Behavioral: eBEfree — Contextual interventions based on promoting acceptance,mindfulness and self-compassion abilities
  Arms: eBEfree

SUMMARY:
The eBEfree project aims at testing the effectiveness of an information and communication technology-based delivery version of BEfree in individuals with obesity and Binge Eating Disorder (BED). BED is a serious public health concern, given its prevalence, psychiatric comorbidity and association with obesity, which is currently a major health and economic challenge of epidemic proportions. BED affects obesity onset, maintenance and treatment. BEfree is a 12-session face-to-face group intervention for BED, developed by the current project research team, that integrates mindfulness, compassion, and values. BEfree was found to be effective in treating BED and in improving psychological adjustment. ICT-based interventions are a cost-effective form of treatment delivery that may increase treatment accessibility for individuals with BED and obesity. This project will directly contribute to the treatment of these conditions and improvement of health services at regional and national levels.

DETAILED DESCRIPTION:
The current project aims at developing a mobile-app adapted version of BEfree - eBEfree - as well as test the efficacy of this ICT-delivery version in a sample of participants with obesity and BED. The specific objectives of the project are:

1. Develop an ICT-delivery version of BEfree: eBEfree.
2. Examine the effectiveness of the ICT-delivery version eBEfree.
3. Test the stability of the outcomes over 6 months.
4. Compare the effectiveness of the eBEfree and the face-to-face version of BEfree.
5. Analyse eBEfree cost-effectiveness.

A detailed description of the aims of the project are presented below.

1. Developing the ICT-delivery version of BEfree - eBEfree. This toolkit will be developed based on the original manual of the face-to-face version of BEfree and will include the tools targeted in BEfree to support participants in reducing BE symptomatology and improve psychological well-being. These tools will cover three main areas:

   i) Mindfulness skills to promote adaptive emotion regulation and improve eating behaviour regulation; ii) Compassion skills to promote motivation that supports sustained adaptive behaviour regulation.

   iii) The development of psychological flexibility and the promotion of values-based living; The techniques of each area will be implemented sequentially in a portfolio of ICT-enabled tools, including a platform with multimedia resources (e.g. videos of sessions) and mobile applications to promote the engagement of users. User evaluation of the platform will be measured using data collected by the mobile application (using metrics like usage time, sessions attended, among others) and through the intervention feedback questionnaire.
2. Examining the effectiveness of the ICT-delivery version eBEfree, through a 2 x 2 factorial Randomized Clinical Trial (RCT) in 70 participants: eBEfree intervention vs. Waiting List Condition (WLC). Primary outcomes are: reductions in BE symptoms and other disordered eating and body image symptoms. Secondary outcomes: Weight loss outcomes; reductions in depressive symptoms and improvements in wellbeing. Mediators of the effectiveness of the ICT-delivery version eBEfree: increases in self-compassion, mindfulness, engagement with valued living, body image psychological flexibility; and decreases in shame, self-criticism and body image-cognitive fusion. Moderators of the intervention: eBEfree engagement (i.e., frequency of mindfulness and compassion meditation practices and daily tasks).
3. Examining the stability of the outcomes measured at 3 and 6 months.
4. Comparing the effectiveness of the eBEfree and the face-to-face version of BEfree, through a 2 x 2 factorial nonrandomized controlled intervention. This aim will be achieved by comparing results from participants who complete the eBEfree intervention and data obtained in the original project BEfree (PTDC/MHC-PCL/4923/2012.).
5. Analysing the cost-effectiveness of the eBEfree by comparing intervention formats: TAU for BED in patients with obesity vs. BEfree, and BEfree vs. eBEfree.

The eBEfree toolkit will include the same components as the original BEfree intervention organized in sequential modules, that will provide psychoeducation of the maintenance cycle of BE, will introduce compassion and mindfulness practices, and will promote psychological flexibility and engagement in values-based actions. A detailed description of each module is provided in Pinto-Gouveia et al. (2016).

The eBEfree will emphasize experiential mindfulness and compassion practices, and daily self-monitoring (i.e., eating behaviour, physical activity). To maximize adherence weekly emails will be sent to participants to prompt engagement with the platform. EBEfree will also include a web-based discussion forum to promote group support and discussion.

Participants Inclusion criteria: a) age: 18-55; b) overweight and obesity (IMC ≥ 25 using a Body Mass Analyzer TANITA-SC-330); c) BED (confirmed through the Eating Disorder Examination 17.0D; d) access to smartphone and willingness to use it regularly (at least once a week).

Exclusion criteria: a) undergoing any other form of psychological intervention for BED or having attended the face-to-face BEfree; b) severe psychiatric problem (e.g., major depression; psychotic illness; bipolar disorder, assessed through a semi-structured interview using DSM-5 criteria).

Results from G*Power calculations for within-group repeated measures analysis, assuming a p value = 0.05, an effect size of f = 0.5, with a statistical power of 0.95, recommend a sample size of 54. Assuming a 20-30% drop-out rate, the minimum sample will be N = 70.

Procedure The sample will be recruited through the dissemination of the study in public health services in the central region of Portugal covered by the Health Centre Regional Administration [Administração Regional de Saúde do Centro - ARSC, IP], a key partner of the project. The study will also be disseminated by the Association of obese and ex-obese patients of Portugal (Associação de Doentes Obesos e Ex-obesos de Portugal, ADEXO) among its members and through its website, which has ≅ 300 daily visits. ADEXO is a nation-wide organization, that promotes the treatment and prevention of obesity. The study will also be advertised in national media outlets.

The advertisement will include a brief description of the project and RT contacts. After contacting the RT, participants will be required to provide informed consent and will be sent a link (through QRCode in flyers or other means) to the eBEfree platform for an online questionnaire to assess eligibility criteria in a first screening phase: age (18-55), self-reported weight status; BE symptomatology (using the Binge Eating Scale cut-off score of > 17); severe depressive symptomatology (using the Beck Depression Inventory cut-off score of > 30); access to smartphone and willingness to use it. If these initial eligibility criteria are met, an individual face-to-face meeting (in the research unit CINEICC), will be scheduled to assess the inclusion criteria described above. Those who meet all inclusion will answer to a set of self-report online questionnaires (3 to 10 presented below) and will be randomly assigned to one of two conditions: eBEfree or WLC. Participants´ responses will be directly sent to a data hub that only the RT will have access to. Those who met criteria for an excluding psychiatric condition will be advised to contact mental health services indicated by the RT. Participants allocated to the eBEfree condition will have access to the eBEfree platform and will be invited to complete eBEfree over the following 12 weeks. After completing the programme participants will be asked to attend an individual face-to-face post intervention assessment where they will be assessed through the EDE 16.0D and the same set of online self-report questionnaires and a post-intervention qualitative feedback questionnaire. Engagement with the online platform data (e.g., practice frequency) will be recorded in the data hub over the 12 weeks of programme completion. Follow-up assessments through online self-report measures (1-10 and self-reported weight) will be conducted at 3 and 6 months.

Participants in the WLC will also complete all assessments and afterwards will be given the opportunity to complete the eBEfree.

ELIGIBILITY:
Inclusion Criteria:

* overweight and obesity (IMC ≥ 25 using a Body Mass Analyzer TANITA-SC-330);
* BED (confirmed through the Eating Disorder Examination 17.0D;
* Access to smartphone and willingness to use it regularly (at least once a week).

Exclusion Criteria:

* undergoing any other form of psychological intervention for BED or having attended the face-to-face BEfree;
* severe psychiatric problem (e.g., major depression; psychotic illness; bipolar disorder, assessed through a semi-structured interview using DSM-5 criteria).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-14 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Reductions in BE symptoms and other disordered eating and body image symptoms | 9 months (from baseline to 6 months follow-up)
  Assessed by EDE interview
Reductions in BE symptoms and other disordered eating and body image symptoms | 9 months (from baseline to 6 months follow-up)
  Assessed by Binge Eating Scale

SECONDARY OUTCOMES:
Weight loss | 9 months (from baseline to 6 months follow-up)
  Measured with a Body Composition Analyzer (Tanita TBF-300)
Reductions in depressive symptoms | 9 months (from baseline to 6 months follow-up)
  Assessed by BDI-II. Beck Depression Inventory-I (Beck, Ward, Mendelson, Mock, & Erbaugh, 1961; Portuguese version by Vaz Serra & Pio Abreu, 1973) is a well-known 21-items questionnaire that measures current depressive symptoms. The Portuguese version shows similar psychometric properties. In the current study, Beck Depression Inventory-I presented an internal consistency of α = .92.
Increasing well-being | 9 months (from baseline to 6 months follow-up)
  Assessed by Obesity Related Wellbeing.Obesity-Related Well-Being Questionnaire (Mannucci, et al., 1999; Silva, Ribeiro, & Cardoso, 2008) is a self-report questionnaire that assesses obesity-related quality of life (QoL), in which higher scores indicate diminished obesity-related QoL. Obesity-Related Well-Being Questionnaire-97 presents good internal consistencies both the original and the Portuguese versions (α = .83 and α = .85 respectively). This study found an α = .86.

OTHER OUTCOMES:
Increase in self-compassion | 9 months (from baseline to 6 months follow-up)
  Assessed by Self-Compassion Scale. Self-Compassion Scale (Neff, 2003; Portuguese version by Castilho, Pinto-Gouveia, & Duarte, 2015) comprises 26 items instrument. Self-Compassion Scale may be used as a two-factor structure: one factor that assess self-compassion attitude and one factor of a self-criticism attitude. Previous studies found adequate model fit and good internal consistency (α = .91 for self-compassion and α = .89 for self-criticism; Costa, Marôco, Pinto-Gouveia, Ferreira, & Castilho, 2015). The current study presented good internal consistencies for both the self-compassion factor (α = .93) and the self-criticism factor (α = .91).
Increase in mindfulness | 9 months (from baseline to 6 months follow-up)
  Assessed by Five Facet Mindfulness Questionnaire. Five Facet Mindfulness Questionnaire-15 (Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006; Portuguese version by Gregório, 2015) is the shorter version of the original 39 items questionnaire that measures the dispositional and multifaceted mindfulness characteristics. Five Facet Mindfulness Questionnaire-15 presents the same five-factor structure as the original version, as well as good internal consistency (ranging from .65 to .86). In the current study, the internal consistencies of the subscales were observing (α = .51), describing (α = .79), act with awareness (α = .50), nonjudgement (α = .68), nonreacting (α = .21). The total scale presented an acceptable internal consistency (α = .70).
Increase in engagement with valued living | 9 months (from baseline to 6 months follow-up)
  Assessed by Engaged Living Scale. Engaged Living Scale (Trompetter et al., 2013) is a self-report measure developed to assess engagement with values-driven behaviour. Recently, a 9-item version of Engaged Living Scale has been used, showing good internal consistency (α = .88; Trindade et al., 2015). The current study found similar internal consistency (α = .82).
Increase in body image psychological flexibility | 9 months (from baseline to 6 months follow-up)
  Assessed by Acceptance and Action Questionnaire - Body Image. BI-AAQ is a 12-item questionnaire designed to measure body image inflexibility (i.e., the ability to accept and experience perceptions, thoughts, beliefs, and feelings relative to one's body without attempting to change their intensity, frequency, or form). This one-dimensional measure has shown good internal consistencies both in the original study (α = .93), and in the Portuguese validation study (α = .95). Also, BI-AAQ discriminates individuals with eating disorders from healthy participants.
Decrease in shame | 9 months (from baseline to 6 months follow-up)
  Assessed by Other as Shamer Scale. Other as Shamer Scale (Goss, Gilbert, & Allan, 1994; Matos, Pinto-Gouveia, Gilbert, Duarte, & Figueiredo, 2015) is an 18-item scale designed to assess individual's perception of being negatively evaluated by others. Other as Shamer Scale has been consistently showing high internal consistency, both in clinical and nonclinical samples (α = .96 and .92, respectively; Goss et al., 1994). In the current study, the scale's internal consistency was α = .94.
Decrease in self-criticism | 9 months (from baseline to 6 months follow-up)
  Assessed by Forms of Self-Criticizing and Reassuring Scale. Forms of Self-Criticising/Attacking & Self-Reassuring Scale (Gilbert et al., 2004) is a 22-item self-report measure of forms of self-criticism (inadequate-self, which focuses on a sense of personal inadequacy ('I am easily disappointed with myself'), and hated-self, which measures the desire to hurt or persecute the self ('I call myself names')) and the ability to self-reassure when things go wrong ('I find it easy to forgive myself'). Cronbach's alphas in non-clinical samples ranged from .89 to .91 for inadequate-self, .82 to .89 for hated-self and .82 to .88 for reassured-self. In clinical samples, Cronbach's alphas ranged from .87 to .89 for inadequate-self, .83 to .86 for hated-self and .85 to .87 for reassured-self. This study found internal consistencies of α = .91 for inadequate-self, α = .67 for hated-self and α = .93 for reassured-self.
Decrease in body-image cognitive fusion | 9 months (from baseline to 6 months follow-up)
  Assessed by Cognitive Fusion Questionnaire - Body Image. Cognitive Fusion Questionnaire-Body Image (Ferreira, Trindade, Duarte, & Pinto-Gouveia, 2015) is a 10-item self-reported questionnaire based on the original Cognitive Fusion Questionnaire (Gillanders et al., 2014). The original study presented good internal consistency, retest reliability, discriminant, and convergent and divergent validities (Trindade, Ferreira, Pinto-Gouveia, & Nooren, 2015). The current study found an internal consistency of α = .95.

CONTACTS AND LOCATIONS:
Overall Officials: José Augusto Pinto Gouveia, PhD, Principal Investigator — University of Coimbra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinto-Gouveia J, Carvalho SA, Palmeira L, Castilho P, Duarte C, Ferreira C, Duarte J, Cunha M, Matos M, Costa J. Incorporating psychoeducation, mindfulness and self-compassion in a new programme for binge eating (BEfree): Exploring processes of change. J Health Psychol. 2019 Mar;24(4):466-479. doi: 10.1177/1359105316676628. Epub 2016 Nov 15. PMID 27852886
- [Background] Pinto-Gouveia J, Carvalho SA, Palmeira L, Castilho P, Duarte C, Ferreira C, Duarte J, Cunha M, Matos M, Costa J. BEfree: A new psychological program for binge eating that integrates psychoeducation, mindfulness, and compassion. Clin Psychol Psychother. 2017 Sep;24(5):1090-1098. doi: 10.1002/cpp.2072. Epub 2017 Jan 25. PMID 28124451
- [Derived] Senra H, Duarte C, Carvalho SA, Simoes L, Ferreira C, Palmeira L, Matos M, Cunha M, Castilho P, Sousa B, Cordeiro L, Pinto-Gouveia J. eBEfree: Combining Psychoeducation, Mindfulness, and Self-Compassion in an App-Based Psychological Intervention to Manage Binge-Eating Symptoms: A Randomized Controlled Trial. Int J Eat Disord. 2025 Jul;58(7):1199-1218. doi: 10.1002/eat.24432. Epub 2025 Mar 29. PMID 40156378